CLINICAL TRIAL: NCT02502799
Title: Intervention for Teens With ADHD and Substance Use
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA034731
Record Dates: First submitted 2015-07-15; First posted 2015-07-20 (Estimated); Results first posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2022-12

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Continued Monitoring and Assessment (Active Comparator): All participants will receive 5 sessions of BEI. Non-responders will then be randomized to one of three conditions. Participants randomized to the continued monitoring and assessment arm will receive no additional intervention. Primary and secondary outcomes will be monitored.
  Interventions: Behavioral: Brief Early Intervention
- PT with ACBT (Active Comparator): All participants will receive 5 sessions of BEI. Non-responders will then be randomized to one of three conditions. For participants randomized to the PT with ACBT arm, parents will participate in behavioral parent training (PT) and adolescents will participate in cognitive behavioral therapy to reduce substance use (CBT).
  Interventions: Behavioral: Brief Early Intervention; Behavioral: Parent Training with Adolescent Cognitive Behavioral Therapy
- PT with ACBT and Methylphenidate (Active Comparator): All participants will receive 5 sessions of BEI. Non-responders will then be randomized to one of three conditions. For participants randomized to the PT with ACBT and Methylphenidate arm, parents will participate in behavioral parent training (PT) and adolescents will participate in cognitive behavioral therapy to reduce substance use (ACBT). Adolescents will also receive methylphenidate.
  Interventions: Behavioral: Brief Early Intervention; Behavioral: Parent Training with Adolescent Cognitive Behavioral Therapy; Drug: Methylphenidate

INTERVENTIONS:
Behavioral: Brief Early Intervention — Adolescents receive 5 individual sessions designed to strengthen the following skills: problem-solving, resisting peer pressure, and coping with emotions. Parents join portions of 3 sessions.
  Other Names: BEI, Teen Intervene
Behavioral: Parent Training with Adolescent Cognitive Behavioral Therapy — Participants receive 12 family sessions with individual adolescent, parent, and joint adolescent and parent time. Includes additional parent training in behavioral modification, adolescent and parent contracting, and adolescent decision-making skills.
  Arms: PT with ACBT; PT with ACBT and Methylphenidate
Drug: Methylphenidate — Adolescents will receive methylphenidate.
  Other Names: Concerta
  Arms: PT with ACBT and Methylphenidate

SUMMARY:
Individuals with ADHD are at markedly high risk for increased substance use and Substance Use Disorder (SUD). Given the strong evidence for the negative trajectory of individuals with co-occurring ADHD and substance use initiation, the goal of this study is to conduct a controlled examination of a brief, early intervention (BEI) for substance modified for adolescents with ADHD. Importantly, this intervention will address individuals who are at risk for problems with substance use, but do not yet meet criteria for severe SUD.

Although brief interventions have been found to be effective in other populations, their efficacy in an ADHD population with emerging risk for substance use problems remains uninvestigated. This study aims to understand why some adolescents with ADHD and elevated risk for SUD respond to (BEI) and others do not. The investigators will test whether situational and individual characteristics predict substance use development and response to treatment. Further, this study will assess which types of additional treatment are most effective for youth who do not respond to the initial BEI. It is hypothesized that rates of adolescent substance use will be lower among adolescents who participate in study treatments.

DETAILED DESCRIPTION:
The goal of this study is to evaluate the efficacy of a brief early intervention (BEI) for reducing early alcohol and marijuana use in a group of 300 adolescents (age 12-16) with ADHD. All adolescents will receive the BEI based on the Teen Intervene program with the addition of enhanced decision making skills. Due to the existing support for the intervention and concern for randomizing families with adolescents at risk for worsening substance use outcomes into a control (no treatment) condition for one to two years, no control condition is used in the current design at the first level of intervention. Similarly, due to the time required to see a potential effect of the treatment (6 months post-brief intervention), a wait-list control condition was not considered.

Adolescents will be evaluated for treatment non-response at 6, 9, 12, 15, and 18 months post-treatment. Non-response is defined as non-normative use of alcohol, marijuana, or other drugs during the past 90 days. Tobacco products are excluded from consideration. Adolescents who demonstrate non-response to the initial BEI at any of the follow-up assessments will be randomized to one of the following conditions: 1) Continued monitoring of substance use with no additional treatment 2) Parent training and adolescent cognitive behavioral therapy (PT/ACBT) 3) PT/ACBT plus concurrent stimulant medication (PT/ACBT + MED). Participants who are randomized will be assessed at 6 months post-treatment and again one year later. The difference in days of substance use at the follow-up assessments among the three conditions will inform which type of intervention is best for youth who do not respond to the initial BEI.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ADHD
* At elevated risk for substance use problems as evidenced by at least one general risk factor (e.g., elevated symptoms of ODD or CD, elevated conflict with parents, low parental monitoring, or academic failure) and at least one substance use specific risk factor (e.g., non-normative use of alcohol or other drugs, use of cigarettes or e-cigarettes, parental substance use problems, family history of substance use problems, peer or sibling substance use).

Exclusion Criteria:

* IQ < 80
* Current substance use disorder meeting DSM-IV criteria for the severe qualifier
* Psychotropic medications for ADHD or any other condition
* Active medical conditions that could be worsened by stimulants unless approved for participation by the treating physician
* Diagnosis of bipolar disorder, schizophrenia, and/or other psychotic disorder
* Diagnosis of autism spectrum disorder (ASD) with a severity level of 2 or 3 or significant intellectual or language impairment

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 158 (Actual)
Dates: Start 2015-07; Primary Completion 2021-08 (Actual); Study Completion 2021-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William E Pelham, PHD, Principal Investigator — Florida International University
Locations (1):
- Florida International University Center for Children and Families, Miami, Florida, United States

REFERENCES:
- [Background] Winters KC, Leitten W. Brief intervention for drug-abusing adolescents in a school setting. Psychol Addict Behav. 2007 Jun;21(2):249-54. doi: 10.1037/0893-164X.21.2.249. PMID 17563146

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants received an initial 5-session substance use prevention program. Participants then completed follow-up assessments to determine level of substance use. Participants identified as having non-normative substance use at any follow-up were moved into the second phase of the study and randomly assigned to one of the three treatment groups. Participants who were never identified as having non-normative substance use were considered responders and were not randomized to a treatment arm.
Groups:
- All Participants: All participants for this study were initially assigned to receive the brief 5-session intervention. Six months following completion of that intervention, follow-up assessments took place to assess response to treatment. At that time, participants identified as "Non-responders" to the brief 5-session intervention were randomly assigned to one of three conditions. Participants (n=109) who were identified as "Responders" were never randomized and received no further intervention. The "Responders" also do not have data for phase 2 of this study because they were never randomized to a treatment arm.
Period: Phase 1: Brief Intervention Sessions
Arm/Group | Continued Monitoring and Assessment | PT With ACBT | PT With ACBT and Methylphenidate | All Participants
Started | 0 (This group did not yet exist during Phase 1: Brief Intervention Sessions. Participants were not randomized to a treatment arm until Phase 2: Intervention Phase. Only participants identified as "Non-responders" during Phase 1, continued to Phase 2.) | 0 (This group did not yet exist during Phase 1: Brief Intervention Sessions. Participants were not randomized to a treatment arm until Phase 2: Intervention Phase. Only participants identified as "Non-responders" during Phase 1, continued to Phase 2.) | 0 (This group did not yet exist during Phase 1: Brief Intervention Sessions. Participants were not randomized to a treatment arm until Phase 2: Intervention Phase. Only participants identified as "Non-responders" during Phase 1, continued to Phase 2.) | 158
Completed | 0 | 0 | 0 | 141
Not Completed | 0 | 0 | 0 | 17
Not completed — Lost to Follow-up | 0 | 0 | 0 | 12
Not completed — Early termination of study | 0 | 0 | 0 | 5
Period: Phase 2: Intervention Phase
Arm/Group | Continued Monitoring and Assessment | PT With ACBT | PT With ACBT and Methylphenidate | All Participants
Started | 16 | 17 | 16 | 0 (Only those participants identified as "Non-responders" during Phase 1 continued to Phase 2 of this study and were randomized to one of the three arms: 1) Continued Monitoring and Assessment; 2) PT with ACBT; 3) PT with ACBT and Methylphenidate)
Completed | 6 | 6 | 7 | 0
Not Completed | 10 | 11 | 9 | 0
Not completed — Lost to Follow-up | 3 | 4 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 3 | 0
Not completed — Study terminated prior to completion | 4 | 5 | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Responders (Never Randomized): These participants received the 5 sessions of BEI; however, were never identified as non-responders to the initial intervention and were never randomized to one of the three treatment groups.
- Total: Total of all reporting groups
Arm/Group | Responders (Never Randomized) | Continued Monitoring and Assessment | PT With ACBT | PT With ACBT and Methylphenidate | Total
Number analyzed (Participants) | 109 | 16 | 17 | 16 | 158
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.77 (1.38) | 14.63 (1.31) | 14.12 (1.17) | 14.25 (1.44) | 13.94 (1.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 3 | 6 | 5 | 41
  Male | 82 | 13 | 11 | 11 | 117
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 2 | 3 | 1 | 14
  White | 84 | 13 | 13 | 14 | 124
  More than one race | 14 | 0 | 1 | 0 | 15
  Unknown or Not Reported | 3 | 1 | 0 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 109 | 16 | 17 | 16 | 158
Past 90-day alcohol use [Count of Participants; unit: Participants] — Teen self-report of alcohol use during the past 90 days.
  Participants
    No use | 82 | 7 | 9 | 7 | 105
    1-2 Times | 18 | 3 | 7 | 7 | 35
    3-5 Times | 3 | 2 | 1 | 0 | 6
    6-9 Times | 5 | 3 | 0 | 1 | 9
    10-19 Times | 0 | 1 | 0 | 1 | 2
    20-39 Times | 1 | 0 | 0 | 0 | 1
    40 Times or More | 0 | 0 | 0 | 0 | 0
Past 90-day marijuana use [Count of Participants; unit: Participants] — Teen self-report of frequency of marijuana use in the past 90 days
  Participants
    No Use | 101 | 6 | 12 | 11 | 130
    1-2 Times | 1 | 2 | 2 | 3 | 8
    3-5 Times | 4 | 2 | 2 | 0 | 8
    6-9 Times | 0 | 3 | 0 | 0 | 3
    10-19 Times | 2 | 1 | 1 | 1 | 5
    20-39 Times | 1 | 1 | 0 | 1 | 3
    40 Times or More | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Past 90-day Alcohol Use
Description: Teen self-report of substance use during the past 90 days
Time Frame: Assessed at 6 months after randomization to treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Continued Monitoring and Assessment | PT With ACBT | PT With ACBT and Methylphenidate
Number analyzed (Participants) | 16 | 17 | 16
Participants
  Missing data on this measure | 6 | 13 | 8
  No alcohol use | 3 | 1 | 1
  Used alcohol 1-2 times | 2 | 3 | 3
  Used alcohol 3-5 times | 3 | 0 | 2
  Used alcohol 6-9 times | 2 | 0 | 1
  Used alcohol 10-19 times | 0 | 0 | 0
  Used alcohol 20-39 times | 0 | 0 | 1
  Used alcohol 40 times or more | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Evidence of Illicit Substances in Urine Screen
Description: Urine analysis indicates presence of illicit substance(s)
Time Frame: Assessed at 6 months after randomization to treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Continued Monitoring and Assessment | PT With ACBT | PT With ACBT and Methylphenidate
Number analyzed (Participants) | 16 | 17 | 16
Participants
  Missing data on this measure | 8 | 13 | 8
  Positive for at least one substance | 3 | 4 | 5
  Negative for all substances | 5 | 0 | 3

3. Secondary Outcome: Mean Youth-Report of Parent-adolescent Conflict
Description: Youth report of conflict with parents on the Conflict Behavior Questionnaire. Higher scores reflect higher parent teen conflict. Total score equals the average across item scores (ranging 1 to 5).
Time Frame: Assessed at 6 months after randomization to treatment
Population: Analysis population includes all participants with complete data on this measure at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Continued Monitoring and Assessment | PT With ACBT | PT With ACBT and Methylphenidate
Number analyzed (Participants) | 6 | 2 | 8
score on a scale | 3.14 (0.11) | 3.15 (0) | 3.00 (0.21)

4. Secondary Outcome: Mean Youth Self-Report of Disruptive Behaviors
Description: Adolescent disruptive behaviors as measured by adolescent self-report and parent report on the Deviant Behavior Scale. Total scores on this measure reflect the average item rating across all items. Scores range from zero to 20 with higher scores reflecting self-report of engaging in more frequent deviant behaviors.
Time Frame: Assessed at 6 months after randomization to treatment
Population: Analysis population includes all participants with complete data on this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Continued Monitoring and Assessment | PT With ACBT | PT With ACBT and Methylphenidate
Number analyzed (Participants) | 10 | 4 | 8
score on a scale | .090 (.166) | .025 (.050) | .100 (.185)

5. Secondary Outcome: Mean Youth Self-Report of Likelihood of Future Substance Use
Description: Youth self-report of likelihood of future substance use during the next year. Score reflects participant report of likelihood of using substances over the next year on a scale from 0 (Definitely will not use) to 10 (Definitely will use).
Time Frame: Assessed at 6 months after randomization to treatment
Population: Analysis population includes all participants with complete data on this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Continued Monitoring and Assessment | PT With ACBT | PT With ACBT and Methylphenidate
Number analyzed (Participants) | 10 | 4 | 8
score on a scale | 5.14 (2.73) | 4.33 (3.06) | 6.00 (1.00)

6. Secondary Outcome: Mean Youth Self-Report of Functional Impairment
Description: Level of impairment experienced across multiple domains of functioning (e.g., at school, at home, with peers) as measured by adolescent self-report on the Impairment Rating Scale. Total score is the mean item rating on a scale from 0 (No problem) to 6 (Extreme problem). Higher scores are indicative of greater impairment.
Time Frame: Assessed at 6 months after randomization to treatment
Population: Analysis population includes all participants with complete data on this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Continued Monitoring and Assessment | PT With ACBT | PT With ACBT and Methylphenidate
Number analyzed (Participants) | 10 | 4 | 8
score on a scale | 1.43 (1.15) | 1.6 (1.74) | 1.91 (.83)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the duration of participation in the study, which could be up to 24 months.
Description: Participants were interviewed about potential adverse events at each follow-up assessment point. Additionally, participants were instructed to notify the investigators in the event of an adverse event between assessment points. Participants identified as "Responders (Never Randomized)" were never randomized to a treatment arm and are therefore not included in adverse event reporting.
Groups:
- Continued Monitoring and Assessment: All participants will receive 5 sessions of BEI. Non-responders will then be randomized to one of three conditions. Participants randomized to the continued monitoring and assessment arm will receive no additional intervention. Primary and secondary outcomes will be monitored.
  Brief Early Intervention: Adolescents receive 5 individual sessions designed to strengthen the following skills: problem-solving, resisting peer pressure, and coping with emotions. Parents join portions of 3 sessions.
  Adverse events for this group represent those report during Phase 2: Intervention Phase.
- PT With ACBT: All participants will receive 5 sessions of BEI. Non-responders will then be randomized to one of three conditions. For participants randomized to the PT with ACBT arm, parents will participate in behavioral parent training (PT) and adolescents will participate in cognitive behavioral therapy to reduce substance use (CBT).
  Brief Early Intervention: Adolescents receive 5 individual sessions designed to strengthen the following skills: problem-solving, resisting peer pressure, and coping with emotions. Parents join portions of 3 sessions.
  Parent Training with Adolescent Cognitive Behavioral Therapy: Participants receive 12 family sessions with individual adolescent, parent, and joint adolescent and parent time. Includes additional parent training in behavioral modification, adolescent and parent contracting, and adolescent decision-making skills.
  Adverse events for this group represent those report during Phase 2: Intervention Phase.
- PT With ACBT and Methylphenidate: All participants will receive 5 sessions of BEI. Non-responders will then be randomized to one of three conditions. For participants randomized to the PT with ACBT and Methylphenidate arm, parents will participate in behavioral parent training (PT) and adolescents will participate in cognitive behavioral therapy to reduce substance use (ACBT). Adolescents will also receive methylphenidate.
  Brief Early Intervention: Adolescents receive 5 individual sessions designed to strengthen the following skills: problem-solving, resisting peer pressure, and coping with emotions. Parents join portions of 3 sessions.
  Parent Training with Adolescent Cognitive Behavioral Therapy: Participants receive 12 family sessions with individual adolescent, parent, and joint adolescent and parent time. Includes additional parent training in behavioral modification, adolescent and parent contracting, and adolescent decision-making skills.
  Methylphenidate: Adolescents will receive methylphenidate.
  Adverse events for this group represent those report during Phase 2: Intervention Phase.
- All Participants: All participants for this study were initially assigned to receive the brief 5-session intervention. Six months following completion of that intervention, follow-up assessments took place to assess response to treatment.
  Adverse events reported below reflect those reported for participants during Phase 1: Brief Intervention.
Arm/Group | Continued Monitoring and Assessment | PT With ACBT | PT With ACBT and Methylphenidate | All Participants
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17 | 0/16 | 0/158
Serious Adverse Events (participants affected / at risk) | 0/16 | 1/17 | 1/16 | 0/158
Other Adverse Events (participants affected / at risk) | 0/16 | 0/17 | 0/16 | 0/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continued Monitoring and Assessment (N=16) | PT With ACBT (N=17) | PT With ACBT and Methylphenidate (N=16) | All Participants (N=158)
Admitted to in-patient psychiatric unit (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | NA — Participant admitted to in-patient psychiatric unit; however, hospitalization was not related to participation in the study.

LIMITATIONS AND CAVEATS:
Enrollment in this study fell well short of the planned 300 participants, despite substantial efforts to increase enrollment over the life of the project, and the study was terminated prior to reaching the planned enrollment target. As a result, the number of participants randomized to treatment condition was insufficient to conduct planned analyses. Furthermore, of those participants randomized, many refused assigned treatments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-07-16): https://cdn.clinicaltrials.gov/large-docs/99/NCT02502799/Prot_SAP_ICF_000.pdf